CLINICAL TRIAL: NCT07340697
Title: An Open-Label Clinical Study to Evaluate the Safety and Effect of RLS-1496 Topical Cream for the Treatment of Actinic Keratosis
Brief Title: Evaluate RLS-1496 Topical Cream for Actinic Keratosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rubedo Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLS-1496-102
Record Dates: First submitted 2026-01-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Single Arm (Experimental): Bilateral Comparison: Active versus Untreated Control
  Interventions: Drug: RLS-1496 1.0% cream

INTERVENTIONS:
Drug: RLS-1496 1.0% cream — Topical cream to be applied to lesions and peri-lesional skin.

SUMMARY:
This clinical trial will assess the safety and tolerability of topical application of RLS-1496 cream to lesions and adjacent skin on the left forearm of adults with actinic keratoses (AK) on the arms. The right forearm will remain untreated as a control. The therapeutic objective of topical treatment with RLS-1496 cream is to clear or decrease the number of AK in the treated area, per lesion counts performed by the Investigator.

The main questions it aims to answer are:

* Is it safe to apply topical RLS-1496 cream to treat AK once daily for 28 days?
* Does topical RLS-1496 lower the number of AKs or eliminate AKs in a treated area when applied once daily for 28 days?

Researchers will compare results on the left (treated with RLS-1496) and right (no treatment) forearm.

Participants will apply RLS-1496 to an identified area on the left forearm once each day for 28 days and have intermittent clinic visits to examine the arms and have the AK lesions counted until 28 days after the last application of RLS-1496. Participants will also have small skin biopsies on the arms.

DETAILED DESCRIPTION:
This open-label study is designed to assess the safety, tolerability, and clinical effects, and pharmacodynamic effects of topically applied RLS-1496 1.0% cream for the treatment of AK lesions and perilesional skin on the left dorsal forearm of adults. The right dorsal forearm will remain untreated as a control.

Eligible patients will apply study drug under the supervision of the study staff to the designated affected area on the left dorsal forearm on Day 1 and will be instructed to apply at home starting on Day 2 and each evening thereafter for a total of 28 applications. Patients will be followed for 28 days after the last application of study drug.

Safety evaluations will include treatment-emergent adverse events (TEAEs), physical examinations, vital signs, local tolerability assessments, and clinical laboratory assessments.

Clinical assessments of treatment effect will be evaluated at each designated treatment and control area. Local tolerability will be assessed. The Investigator will count discrete AK lesions within the designated treatment and control areas.

Additional assessments will include selected disease-specific biomarkers and markers for target engagement, and senescence in the skin (biopsy and tape stripping), and in the blood.

Following a screening period of up to 28 days, eligible participants will be dosed through Day 28 and followed for an additional 28 days. The predicted maximum duration of study participation, including the screening period, is 85 days.

Approximately 24 patients will be enrolled in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* area on each dorsal forearm with 4-12 clinically typical, discrete and visibly evident AK lesions within a 25-100 cm2 area
* willing to comply with the study requirements, including refraining from use of medications or other treatments for the skin disease (including sun and ultraviolet light exposure), and is able to reliably apply topical medications

Key Exclusion Criteria:

* significant skin disease other than AK which may interfere with interpretation of clinical findings
* atypical or rapidly changing AK lesions at the intended treatment and control area (including cutaneous horn, hyperkeratotic, hypertrophic lesions)
* clinically relevant co-morbid medical conditions or findings on physical examination or in laboratory analyses
* known or suspected pregnancy or lactation (female patients), or planned pregnancy (female and female partners of male patients)
* treatment with 5-fluorouracil (5-FU), tirbanibulin, imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for AK within the intended treatment and control area or within 2 inches (or 5 cm) of the treatment and control area, within 28 days prior to Screening and Day 1visit
* treatment with cosmetic or therapeutic procedures (eg, use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing), use of acid-containing therapeutic products (eg, salicylic acid or fruit acids, such as alpha and beta-hydroxyl acids and glycolic acids), topical retinoids, light chemical peels, topical steroids, artificial tanners, or other topical medicinals (non-medicated and non-irritating lotions or creams are permitted) within the intended treatment and control area or within 2 inches (or 5 cm) of the treatment and control area, within 14 days prior to Screening and Day 1 visit
* treatment with immunomodulators (eg, azathioprine), cytotoxic drugs (eg, cyclophosphamide, vinblastine, chlorambucil, methotrexate), interferons/interferon inducers, medications that suppress the immune system (eg, cyclosporine, prednisone, methotrexate, alefacept, infliximab) within 28 days prior to Screening and Day 1 visit
* treatment with systemic retinoids (eg, isotretinoin, acitretin, bexarotene) within 6 months prior to Screening and Day 1 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety of multiple doses of topical RLS-1496 cream | 57 days
  Treatment-emergent adverse events
Proportion of individual AK lesions with complete (100%) clearance | 29 days
  AK lesions with 100% clearance in the treatment and control area at Day 29 (versus pre-dose on Day 1)
Complete (100%) clearance of AK lesions | 29 days
  100% clearance of AK lesions in the treatment and control area at Day 29 (versus pre-dose on Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Director — Acting Chief Medical Officer
Locations (4):
- United States (4):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Schlessinger MD Skin Research Center, Omaha, Nebraska
  - Austin Institute for Clinical Research, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No